CLINICAL TRIAL: NCT04063423
Title: Non- Clinical Coagulation Activation During Hemodialysis: a Cross-sectional Study Evaluating Agreement and Correlation Between Hemodialysis Session Parameters, Biological Markers and Objective Measurements of Hemodialyzers: "NC-coact"
Brief Title: Non- Clinical Coagulation Activation During Hemodialysis
Acronym: NC-Coact
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: UZB-NEF-2018-NC-COACT
Record Dates: First submitted 2019-01-22; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Kidney Diseases; End Stage Renal Disease; Hemodialysis Complication
Keywords: clotting; coagulation
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic; Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hemodialysis study session: * 4h hemodialysis session using standard polysulphone dialyzer and Nikkiso dialysis monitors
  * Minimal dose of unfractionated heparin (UFH) with loading dose 500IE and maintenance 500IE/h, stopped 60 minutes before session end in case of AVF use.
  * Standard bicarbonate-based ultrapure dialysate. Na, K, Ca, bicarbonate concentrations according to the patient's routine dialysis prescription.
  * The blood flow rate maximized as per routine nursing care.
  * Dialysate flow rate fixed at 500 ml/min.
  * Dialysate temperature between 35.5°C and 36.5°C.
  * Ultrafiltration according to patient's dry weight and supported ultrafiltration rate.
  * At the end of the dialysis session the blood will be returned (100ml/min) to the patient.
  Interventions: Procedure: blood sample

INTERVENTIONS:
Procedure: blood sample — Blood sample at start and at the end of the dialysis session; membrane scoring after dialysis; total cell volume measurement of dialyzer after dialysis; micro-CT of dialyzer after dialysis.

SUMMARY:
Every patient included in the study will undergo 1 conventional hemodialysis treatment, ie 1 study visit. During the conventional hemodialysis treatment lasting 4 hours, 2 blood samples will be taken at different time points (5 minutes after dialysis start and 240 minutes after dialysis = at the end of the dialysis session) to evaluate coagulation activation (TAT, PF1+2). Hemodialysis session parameters (arterial and venous pressure, TMP, OCM, BVM and prefilter pressure) will be noted at different time points (T5, T30, T60, T120, T180, T240). After discontinuation of the dialysis session, total cell volume will be measured using the Renatron II system® and the number of open fibers will be determined using micro-CT scanning.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Patients able and agree to provide signed informed consent.

Exclusion Criteria:

* Known allergy for polysulphone dialysis membrane.
* Use of vitamin K antagonists or novel oral anticoagulant therapy.
* Use of chronic heparin treatment, UFH or LMWH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with end stage renal disease treated with hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
TAT | From first hemodialysis study session until interpretation of biological results, up to 6 months
  thrombin antithrombin complex levels (mcg/L). Samples for TAT measurement were taken during the single hemodialysis study treatment. All patients underwent their study treatments between October - December 2018. All analyses were performed in batch in January 2019.
open fibers | From first hemodialysis study session until interpretation of scan results, up to 6 months
  number of open fibers of dialyzer counted after microCT scanning of dialyzer membrane. Dialyzers were collected after the hemodialysis study treatment. All patients underwent their study treatments between October - December 2018. All micro CT scans were performed using the same scanner in Fabruary and March 2019.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: Undecided